CLINICAL TRIAL: NCT01233908
Title: Diagnosis of Posttraumatic Stress Disorder Following Primary Rhegmatogenous Retinal Detachment
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Ido Didi Fabian, MD, Sheba medical center
Other Study IDs: SHEBA-10-7609-DF-CTIL
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Stress Disorders, Post-Traumatic; Retinal Detachment
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PTSD: Patients which underwent surgical repair for primary rhegmatogenous retinal detachment and developed an associated posttraumatic stress disorder
- PTSD - negative: Patients which underwent surgical repair for primary rhegmatogenous retinal detachment and did not develope an associated posttraumatic stress disorder

SUMMARY:
To investigate the prevalence of posttraumatic stress disorder (PTSD) in patients that underwent surgery for primary rhegmatogenous retinal detachment (RRD) and to determine variables associated with the disorder.

Design: Consecutive prospective observational study.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD) is a potentially blinding condition and a common cause of ocular morbidity, with an estimated incidence of 6.3-17.9 per 100,000 of population. 1 Despite contemporary surgical treatments, with nearly 95% of anatomical success, functional results for the repair of primary RRD remain poor, with only 43% achieving a final vision ≥ 20/40 and 21% a visual acuity (VA) < 20/100. 2 Various studies of vision related quality of life after RRD have demonstrated that RRD subjects suffer with substantial impairment of physical, psychological and social functions. 3-6 Mozaffarieh et al. further demonstrated that these subjects suffer of anxiety and depression, with correlation to visual functional status. 7 However, to date, no study have assessed the occurrence of primary RRD as a traumatic event that may trigger an associated distress disorder.

Post traumatic distress disorder (PTSD) is diagnosed after a subject is exposed to an extreme stressor or traumatic event, which resulted with response of fear, helplessness, or horror, and caused typical symptoms of reexperiencing of the event, avoidance of reminders of the event, and increased arousal, for at least one month (Table 1). 8 PTSD was found to occur in the aftermath of external traumas, such as rape, physical assault, combat and natural disasters. 9 However, various illnesses were described as well, as triggering events, after which PTSD developed: myocardial infarction (MI), 10 abortions, 11, 12 cancer, 13 diagnosis of HIV infection, 14 and pulmonary diseases. 15, 16 The burden of PTSD can be high, with inability to work or return to prior levels of functioning. 17, 18 The work impairment associated with PTSD is estimated to result with an annual productivity loss in excess of $3 billion in the US. 19 Furthermore, PTSD was found to have an impact on physical health, with higher rates of cardiovascular and pulmonary illnesses, 20 and with greater utilization of health care services, 21 all together putting the disorder as a major public health problem.

The purpose of our study was to examine whether the occurrence of a primary RRD can give rise to an associated PTSD, to investigate its prevalence and determine variables associated with the disorder.

Methods:

We approached 547 patients with a previous primary RRD, of which 363 (mean age 58 ± 15 years, 64% were men) were enrolled in the study. PTSD was assessed by the Clinician Administered PTSD Scale and the 25-Item National Eye Institute Visual Function Questionnaire (NEI-VFQ-25) was used as a measure of vision-related quality of life. Objective clinical measures were obtained from the patient's medical records. Psychological and ophthalmological variables were compared between PTSD diagnosed patients and a subset of PTSD-negative patients, who served as controls.

ELIGIBILITY:
Inclusion Criteria:

Above 18 years of age, underwent surgical correction for primary rhegmatogenous retinal detachment, follow up of at least 1 month after surgery

Exclusion Criteria:

Poor Hebrew proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for the study were subjects, above 18 years of age, who underwent surgical correction for primary rhegmatogenous retinal detachmentat the Goldschleger Eye Institute, from January 1, 2004 to September 31, 2009, and were followed up for at least 1 month
Sampling Method: Non-Probability Sample
Enrollment: 547 (Actual)
Dates: Start 2010-01; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Diagnosis of posttraumatic stress disorder

CONTACTS AND LOCATIONS:
Overall Officials: Ido Didi Fabian, MD, Study Chair — Chaim Sheba medical center
Locations (1):
- Goldschleger institute of ophthalmology, Sheba medical center, Ramat Gan, Israel

REFERENCES:
- [Background] Mitry D, Charteris DG, Fleck BW, Campbell H, Singh J. The epidemiology of rhegmatogenous retinal detachment: geographical variation and clinical associations. Br J Ophthalmol. 2010 Jun;94(6):678-84. doi: 10.1136/bjo.2009.157727. Epub 2009 Jun 9. PMID 19515646
- [Background] Pastor JC, Fernandez I, Rodriguez de la Rua E, Coco R, Sanabria-Ruiz Colmenares MR, Sanchez-Chicharro D, Martinho R, Ruiz Moreno JM, Garcia Arumi J, Suarez de Figueroa M, Giraldo A, Manzanas L. Surgical outcomes for primary rhegmatogenous retinal detachments in phakic and pseudophakic patients: the Retina 1 Project--report 2. Br J Ophthalmol. 2008 Mar;92(3):378-82. doi: 10.1136/bjo.2007.129437. PMID 18303159
- [Background] Sullivan PM, Luff AJ, Julious SA, Canning CR. Patient satisfaction following vitreoretinal surgery. Eye (Lond). 1993;7 ( Pt 3):433-5. doi: 10.1038/eye.1993.86. PMID 8224301
- [Background] Zou H, Zhang X, Xu X, Liu H. Quality of life in subjects with rhegmatogenous retinal detachment. Ophthalmic Epidemiol. 2008 Jul-Aug;15(4):212-7. doi: 10.1080/09286580701843804. PMID 18780253
- [Background] Globe DR, Levin S, Chang TS, Mackenzie PJ, Azen S. Validity of the SF-12 quality of life instrument in patients with retinal diseases. Ophthalmology. 2002 Oct;109(10):1793-8. doi: 10.1016/s0161-6420(02)01124-7. PMID 12359596
- [Background] Scott IU, Smiddy WE, Feuer W, Merikansky A. Vitreoretinal surgery outcomes: results of a patient satisfaction/functional status survey. Ophthalmology. 1998 May;105(5):795-803. doi: 10.1016/S0161-6420(98)95017-5. PMID 9593378
- [Background] Mozaffarieh M, Sacu S, Benesch T, Wedrich A. Mental health measures of anxiety and depression in patients with retinal detachment. Clin Pract Epidemiol Ment Health. 2007 Jul 19;3:10. doi: 10.1186/1745-0179-3-10. PMID 17640389
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Gander ML, von Kanel R. Myocardial infarction and post-traumatic stress disorder: frequency, outcome, and atherosclerotic mechanisms. Eur J Cardiovasc Prev Rehabil. 2006 Apr;13(2):165-72. doi: 10.1097/01.hjr.0000214606.60995.46. PMID 16575268